CLINICAL TRIAL: NCT00628446
Title: Prevalence and Risk of Coronary Heart Disease as Measured by Coronary Calcium Score Among Individuals With Chronic Traumatic Spinal Cord Injury(SCI): A Pilot Study
Brief Title: Coronary Heart Disease as Measured by Coronary Calcium Score Among Individuals With Chronic Traumatic Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CCS-040
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2015-07

CONDITIONS: Spinal Cord Injuries; Heart Diseases
Keywords: spinal cord injury; Coronary artery calcium; Dyslipidemia
MeSH Terms: conditions — Spinal Cord Injuries; Heart Diseases; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study includes male subjects age 45 to 70, who have sustained a traumatic Spinal Cord Injury (SCI) at least 10 years prior. Subjects will be interviewed for demographic data, including heart disease risk factors. A blood test for cholesterol levels will be drawn. A CT scan of arteries of the heart will be performed to determine the presence of coronary calcium, a marker of subclinical Coronary Heart Disease. Scoring of Coronary Calcium or Coronary Calcium Score (CCS) is automated by the CT scanner. Each subject's Framingham Risk Score will be calculated; This is an individuals 10 year risk of having a Coronary Heart Disease event (significant symptoms). In addition, it will be determined if subjects are being treated for diagnosed dyslipidemia (high cholesterol) according to the National Cholesterol Educational Program (NCEP) guidelines.

The proposed pilot study aims to better understand the problem of Coronary Heart Disease in individuals with Spinal Cord Injury, specifically CCS in SCI, when compared to the general population.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Spinal Cord Injury due to externally inflicted trauma
* > or = 10 years post injury
* American Spinal Injury Association (ASIA) Scale A,B, or C
* 45 to 70 years of age
* Communication and comprehension sufficient for compliance with all testing procedures
* Voluntary informed consent

Exclusion Criteria:

* Spinal Cord Injury of non-traumatic etiology
* Injury < 10 years prior to enrollment
* Known Coronary Heart Disease

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male,Spinal Cord Injuries
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Lieberman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

REFERENCES:
- [Result] Lieberman JA, Hammond FM, Barringer TA, Norton HJ, Goff DC Jr, Bockenek WL, Scelza WM. Comparison of coronary artery calcification scores and National Cholesterol Education program guidelines for coronary heart disease risk assessment and treatment paradigms in individuals with chronic traumatic spinal cord injury. J Spinal Cord Med. 2011;34(2):233-40. doi: 10.1179/107902610X12923394765733. PMID 21675362
- [Result] Lieberman JA, Hammond FM, Barringer TA, Goff DC Jr, Norton HJ, Bockenek WL, Scelza WM. Adherence with the National Cholesterol Education Program guidelines in men with chronic spinal cord injury. J Spinal Cord Med. 2011;34(1):28-34. doi: 10.1179/107902610x12883422813589. PMID 21528624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in 2007 and was completed in 2008. All recruitment was done at the Carolinas Rehabilitation Outpatient SCI clinic
Period: Overall Study
Arm/Group | Study Group
Started | 45
Completed | 38
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Percent Agreement Between Coronary Calcium Score (CCS) and National Cholesterol Education Program (NCEP) Guidelines
Description: Participants were classified as high risk, intermediate high risk, intermediate low risk, and low risk based upon both their CCS and their LDL using NCEP Adult Treatment Panel III Guidelines. Those with CCS >/-400 were considered high risk, CCS=100-399 were intermediate high risk, CCS=1-99 intermediate low risk, and CCS=0 were low risk. The percent agreement between CCS and NCEP Guidelines was calculated by totaling the number of subjects who were classified in the same risk category and dividing by the total number of subjects
Time Frame: During single data collection. Average duration of injury was 24.4 years +/-9.5 years
Measure: Number; unit: percent agreement
Groups:
- Study Group: Cross-sectional study group
Arm/Group | Study Group
Number analyzed (Participants) | 38
percent agreement | 18

2. Secondary Outcome: Adherence to NCEP Criteria
Description: Determine the total percentage of subjects who should be on drug therapy by NCEP criteria and who are on drug therapy who have achieved their treatment goal as defined by NCEP criteria
Time Frame: During single data collection
Population: 38 subjects completed the data collection
Measure: Number; unit: percentage of participants
Arm/Group | Group 1
Number analyzed (Participants) | 38
percentage of participants | 39.5

ADVERSE EVENTS:
Time Frame: September 2007-November 2008
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No